CLINICAL TRIAL: NCT01251523
Title: Improving Asthma Outcomes Through Cultural Competence Training for Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Randall Brown, PI, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R01HL09338601A2
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PACE Plus (Active Comparator): Physicians enrolled in the study will be randomized to one of three arms: Control, PACE intervention or PACE Plus intervention. Their pediatric asthma patients enrolled in the study will follow them into their randomization assignment.
  Interventions: Behavioral: PACE Plus
- PACE (Active Comparator): Physicians enrolled in the study will be randomized to one of three arms: Control, PACE intervention or PACE Plus intervention. Their pediatric asthma patients enrolled in the study will follow them into their randomization assignment.
  Interventions: Behavioral: PACE
- Control (No Intervention): Physicians enrolled in the study will be randomized to one of three arms: Control, PACE intervention or PACE Plus intervention. Their pediatric asthma patients enrolled in the study will follow them into their randomization assignment.

INTERVENTIONS:
Behavioral: PACE — The first intervention to be tested, Physician Asthma Care Education (PACE), is a rigorously evaluated intervention for physicians that has reached hundreds of clinicians across the U.S. and also has been implemented in the United Kingdom and Australia. The efficacy trial of PACE was supported by the National Heart, Lung and Blood Institute and the effectiveness trial by the Robert Wood Johnson Foundation. PACE is now widely available to clinicians, through, among other channels, the National Asthma Education and Prevention Program (NAEPP). It is designed to enhance physician communication, counseling and therapeutics for assisting the general population of children with asthma.
  Other Names: PACE (Physician Asthma Care Education)
  Arms: PACE
Behavioral: PACE Plus — In the PACE PLUS intervention a cultural competence component will be added to the PACE curriculum. The cultural competence component uses mini-lecture, video demonstration (video to be developed as part of this proposal), case studies and self observation tools to present the principles of cultural competence derived from the study of the literature. The component integrates into the skills taught, specific content related to working with African American and Puerto Rican families where a child has asthma.
  Arms: PACE Plus

SUMMARY:
The proposed randomized clinical trial will compare two educational interventions: Physicians Asthma Care Education (PACE) and PACE Plus with 90 physicians in Atlanta and the Bronx and their 1192 patients.

DETAILED DESCRIPTION:
Massive resources are expended every year on cultural competence training for physicians. However no rigorous study that has assessed whether cultural competence training for physicians results in better health outcomes for their patients.

The investigators propose to conduct a randomized clinical trial to compare two interventions. The study will involve three groups. The first, Physician Asthma Care Education (PACE), is a proven program for enhancing communication, therapeutic practice and the ability of physicians to foster effective management of asthma by their patients in general. The second is the PACE program plus skills and concepts considered in the literature essential to culturally competent practice (PACE PLUS). It is designed to give clinicians a higher degree of certainty and confidence in working across cultures. PACE PLUS was specifically developed to enable physicians to understand and overcome potential biases in their interactions with patients whose racial/ethnic identity is different from their own. The third is a control group that will not receive an intervention. Two racial/ethnic groups of patients will be the focus of the research: African American and Latino/Hispanic, specifically, Puerto Rican children with asthma and their parents or caretakers. The proposed study will evaluate the effects of the training for physicians on health outcomes for the children and performance ratings given to the physician by the parent of the child.

The proposed study will address two questions:

1. Does cultural competence training (PACE PLUS) produce better outcomes for minority patients, specifically African American and Puerto Rican children, and their respective parents, than a general communication training program (PACE)?
2. Compared to the control group, is the Physician Asthma Care Education program (PACE), already shown to be effective with the general population of patients, effective when used with minority patients, specifically African American and Puerto Rican children, and their parents?

The study hypothesis is that there will be positive outcomes for patients of physicians in both interventions but better outcomes for those patients whose doctors participate in the cultural competence training (PACE PLUS). That is:

1. PACE PLUS compared to PACE will produce:

   * reductions in children's health care use for asthma
   * improved symptom experience for the children
   * greater parent/caretaker satisfaction with the physician's performance
   * enhanced asthma related quality of life for parents/caretakers of the patients
   * higher levels of confidence and value placed by physicians on skills needed when working cross culturally
   * increased use of National Asthma Education and Prevention Program (NAEPP) recommended therapies by physicians
2. PACE compared to a control group will produce better outcomes on these six dimensions.

ELIGIBILITY:
Inclusion Criteria:

* Physician enrollment criteria are: 1) licensed physician in practice and board certified in pediatrics or family medicine; 2) treating children with asthma; 3) full-time in a practice in Atlanta, GA or New York City, NY; 4) not Latino/Hispanic or African American in ethnicity/race; 5) consenting to participate and 6) will generate a roster of pediatric asthma patients.

The following patient selection criteria will be used.

* The child must: 1) be treated by the participating physician during the study intake period; 2) be between one and 16 years of age; 3) have a diagnosis of asthma made by a physician using the NAEPP Guidelines for the diagnosis of asthma (NHLBI, 2007) (The investigators will not accept alternative descriptions such as reactive airway disease, bronchitis, or wheezy bronchitis. The determination must be asthma); 4) have at least one emergency medical care visit in the previous year (hospitalization, or ED or physician office visit on an emergency basis defined as administration of epinephrine sub-cutaneously or bronchodilators by aerosol); 5) not have other chronic disorders that have pulmonary complications, e.g. sickle cell disease; 6) be of self-identified African American or Latino/Hispanic race/ethnicity.
* In addition, the parent/caretaker must meet the following criteria: 1) be the one usually responsible for the child's car; 2) be of self identified African American or Latino/Hispanic race/ethnicity; 3) have access to a telephone; and 4) consent to participate.

Exclusion Criteria:

* Physicians and patients who cannot meet the above inclusion criteria

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1176 (Actual)
Dates: Start 2010-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Emergency Department Visits - 1st time point | 12 months prior to baseline interview
  The investigators will collect health care utilization data related to the child's asthma. Parents of the pediatric subjects will complete a telephone interview at baseline. During that interview they will be asked to provide information regarding the frequency of asthma related Emergency Department visits (for the child) during the year prior to the baseline interview. A subset of the patients will have their records reviewed at their doctor's office for asthma related ED visits during this time period.
Emergency Department Visits - 2nd time point | Interval between baseline and 9 months
  The investigators will collect health care utilization data on the child subject of this study. Parents of the pediatric patients will be asked during their 9 month follow up telephone interview about the frequency of asthma related ED visits (for the child) during the interval since the baseline interview (baseline - 9 months). In addition, a subset of the patients in the study will have their records reviewed in the clinic for a reporting of asthma related ED visits.
Emergency Department Visits - 3rd time point | interval between 9 month and 18 month telephone interview
  The investigators will collect health care utilization data related to asthma. Parents of the child subjects in the study will be asked during their 18 month telephone interview to recall the frequency of asthma related ED visits for the child in the last year since their 9 month telephone interview. In addition, a subset of children will have their records accessed at their drs office for a reporting of ED visits.

SECONDARY OUTCOMES:
Hospitalizations - first time point | Year prior to baseline interview
  The investigators will ask parents of the child subjects during their baseline telephone interview to provide information on hospitalizations related to asthma in the year prior to their baseline interview. In addition, the investigators will review patient records at the clinic for a subset of the children for hospitalizations during this period.
Hospitalizations - 2nd time point | Interval between baseline and 9 month telephone interview
  The investigators will ask parents of the child subjects during their 9 month telephone interview to provide information on hospitalizations related to asthma in the year between their baseline and 9 month interview. In addition, the investigators will review patient records at the clinic for a subset of the children for hospitalizations during this period.
Hospitalizations - 3rd time point | interval between 9 month and 18 month telephone interview
  The investigators will ask parents of the child subjects during their 18 month telephone interview to provide information on hospitalizations related to asthma in the year between their 9 month and 18 month interview. In addition, the investigators will review patient records at the clinic for a subset of the children for hospitalizations during this period.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Brown, MD, MPH, Principal Investigator — University of Michigan School of Public Health
Locations (1):
- University of Michigan School of Public Health, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Patel MR, Song PXK, Bruzzese JM, Hao W, Evans D, Thomas LJ, Pinkett-Heller M, Meyerson K, Brown RW. Does cross-cultural communication training for physicians improve pediatric asthma outcomes? A randomized trial. J Asthma. 2019 Mar;56(3):273-284. doi: 10.1080/02770903.2018.1455856. Epub 2018 Apr 11. PMID 29641357
- [Derived] Patel MR, Thomas LJ, Hafeez K, Shankin M, Wilkin M, Brown RW. Study protocol for improving asthma outcomes through cross-cultural communication training for physicians: a randomized trial of physician training. BMC Med Educ. 2014 Jun 16;14:118. doi: 10.1186/1472-6920-14-118. PMID 24935221